CLINICAL TRIAL: NCT01912287
Title: GATE: Generalized Anxiety - A Treatment Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: s17-00526; 1R01AT007258-01A1 (NIH); NCT03445143 (obsolete NCT alias)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; GAD; Yoga; CBT
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga (Experimental): The yoga intervention will apply Kundalini Yoga practices as taught by Yogi Bhajan. This is a well-known, accessible style of practice in the U.S. that incorporates all of the traditional components of yoga including physical postures and exercises, breathing techniques, relaxation exercises and meditation practices. It is a safe style of yoga that is registered with the Yoga Alliance that is readily and routinely adapted for therapeutic purposes. The 12-week yoga intervention will consist of 12 group classes and assigned daily home practice led by qualified and certified yoga instructors. Each group yoga session will include physical postures/exercises, breathing techniques, meditation and deep relaxation practice that are all easy to learn and do not require extensive practice or athletic ability to perform.
  Interventions: Behavioral: Yoga
- Cognitive Behavioral Therapy (CBT) (Active Comparator): The 12 session CBT treatment will be based on the standardized protocol developed at one of our centers (CARD) and widely available [88]. This protocol is comprised of four primary treatment modules including cognitive restructuring, progressive muscle relaxation, worry exposures, and in vivo exposure exercises. The initial sessions describe the cognitive behavioral model of worry and GAD. Each session consists of a different "lesson." These lessons initially cover basic information about the nature of the anxiety and worry, the possible function and negative consequences of worrying, the maladaptive and paradoxical effects of attempting to control and suppress one's thoughts, the basic cognitive errors of probability overestimation and catastrophic thinking, adaptive strategies to deal with worries, such as problem solving, worry exposure, which may involve exploring and exposing the patient to negative images and scenarios that might be behind some of the worrisome thoughts.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Stress Education (Sham Comparator): SE will also include 12 weeks of group and home practice sessions. SE will control for attention from instructors, expectancy effects, and group support effects, Stress Education (SE) will be employed as an active control intervention. SE is currently used in NIH-funded protocols at the Benson-Henry Institute for Mind-Body Medicine at MGH. In this condition, participants will be provided with detailed and extensive information about stress and health, but will not receive any CBT, yoga, or other mind-body training techniques.
  Interventions: Behavioral: Stress Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT focused on Generalized Anxiety Disorder (12 sessions)
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Stress Education — Active control group (12 sessions)
  Other Names: SE
  Arms: Stress Education
Behavioral: Yoga — 12 sessions, mindfulness components
  Other Names: Kundalini Yoga
  Arms: Yoga

SUMMARY:
The purpose of this randomized study is to examine the comparative efficacy of yoga, cognitive behavioral therapy, and stress education, a previously employed control condition, for patients with Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
We are currently conducting a treatment study to reduce stress and anxiety in people with generalized anxiety disorder (GAD). This study will not use a medication, but instead will involve weekly stress reduction classes that use different strategies to reduce anxiety. The study involves having a formal psychiatric interview, filling out questionnaires, ECGs, saliva samples, a urine test for drugs of abuse, and study visits over 12 weeks. Each study visit will take a few hours. Qualified participants will be compensated for time and travel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients > 18 years of age with a primary psychiatric diagnosis of generalized anxiety disorder
* Clinical Global Impression-Severity scale (CGI-S) score of 4 or higher
* Off concurrent psychotropic medication for at least 2 weeks prior to initiation of randomized treatment, OR stable on current medication for a minimum of 6 weeks and willing to maintain a stable dose
* Willingness and ability to perform the yoga intervention and to comply with the requirements of the study protocol.
* For women of childbearing potential, willingness to use a reliable form of birth control

Exclusion Criteria:

* Patients unable to understand study procedures and participate in the informed consent process.
* Pregnancy as assessed by pregnancy test at screen or lack of use approved methods birth control for women of childbearing age
* Women who are planning to become pregnant
* Serious medical illness or instability for which hospitalization may be likely within the next year
* Significant current suicidal ideation or suicidal behaviors within the past 6 months (assessed with the Beck Depression Inventory-II [BDI-II])
* History of head trauma causing loss of consciousness, or seizure disorder resulting in ongoing cognitive impairment
* Posttraumatic stress disorder, substance use disorder, eating disorder, or organic mental disorder within the past 6 months
* Lifetime history of psychotic disorder, bipolar disorder, or developmental disorder
* Significant personality dysfunction likely to interfere with study participation (assessed during the clinical interview)
* Prior experience with (more than 5 Yoga classes or CBT sessions within the last 3 years) and/or current practice of mindbody techniques (e.g., yoga, meditation, Tai-Chi, etc) or cognitive behavioral therapy (CBT)
* Concomitant therapy for generalized anxiety disorder (GAD) (any therapy)
* Physical conditions that might cause injury from yoga (pregnancy, physical injuries and musculoskeletal problems)
* Cognitive impairment (MOCA<21)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2013-12; Primary Completion 2019-04-29 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Simon, MD, MSc, Principal Investigator — NYU Langone Health; Stefan G Hofmann, PhD, Principal Investigator — Boston University; Eric Bui, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keltz S, Quintana L, Szuhany KL, Adhikari S, Twi-Yeboah A, Baker AW, Khalsa SBS, Hoge E, Bui E, Hoeppner SS, Rosenfield D, Hofmann SG, Simon NM. Impact of homework engagement on treatment response to group cognitive-behavioral therapy, yoga, and stress education for generalized anxiety disorder. Cogn Behav Ther. 2025 Nov 18:1-12. doi: 10.1080/16506073.2025.2589392. Online ahead of print. PMID 41252645
- [Derived] Hoge EA, Simon NM, Szuhany K, Feldman B, Rosenfield D, Hoeppner S, Jennings E, Khalsa SB, Hofmann SG. Comparing Kundalini Yoga, cognitive behavioral therapy, and stress education for generalized anxiety disorder: Anxiety and depression symptom outcomes. Psychiatry Res. 2023 Sep;327:115362. doi: 10.1016/j.psychres.2023.115362. Epub 2023 Aug 6. PMID 37598625
- [Derived] Szuhany KL, Adhikari S, Chen A, Lubin RE, Jennings E, Rassaby M, Eakley R, Brown ML, Suzuki R, Barthel AL, Rosenfield D, Hoeppner SS, Khalsa SB, Bui E, Hofmann SG, Simon NM. Impact of preference for yoga or cognitive behavioral therapy in patients with generalized anxiety disorder on treatment outcomes and engagement. J Psychiatr Res. 2022 Sep;153:109-115. doi: 10.1016/j.jpsychires.2022.07.008. Epub 2022 Jul 5. PMID 35810600
- [Derived] Simon NM, Hofmann SG, Rosenfield D, Hoeppner SS, Hoge EA, Bui E, Khalsa SBS. Efficacy of Yoga vs Cognitive Behavioral Therapy vs Stress Education for the Treatment of Generalized Anxiety Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Jan 1;78(1):13-20. doi: 10.1001/jamapsychiatry.2020.2496. PMID 32805013

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Therapy (CBT): The 12 session CBT treatment will be based on the standardized protocol developed at one of our centers (CARD) and widely available. This protocol is comprised of four primary treatment modules including cognitive restructuring, progressive muscle relaxation, worry exposures, and in vivo exposure exercises. The initial sessions describe the cognitive behavioral model of worry and GAD. Each session consists of a different "lesson." These lessons initially cover basic information about the nature of the anxiety and worry, the possible function and negative consequences of worrying, the maladaptive and paradoxical effects of attempting to control and suppress one's thoughts, the basic cognitive errors of probability overestimation and catastrophic thinking, adaptive strategies to deal with worries, such as problem solving, worry exposure, which may involve exploring and exposing the patient to negative images and scenarios that might be behind some of the worrisome thoughts.
Period: Overall Study
Arm/Group | Yoga | Cognitive Behavioral Therapy (CBT) | Stress Education
Started | 93 | 90 | 43
Completed | 60 | 67 | 28
Not Completed | 33 | 23 | 15
Not completed — Ineligible | 1 | 0 | 1
Not completed — No-show | 0 | 0 | 1
Not completed — Dissatisfaction with assigned treatment | 4 | 2 | 1
Not completed — Felt treatment no longer needed | 0 | 1 | 0
Not completed — Life circumstances | 4 | 2 | 0
Not completed — Lost Interest | 1 | 0 | 0
Not completed — Uknown reason - subject drop out | 5 | 7 | 3
Not completed — Missed Assesment | 1 | 1 | 1
Not completed — Scheduling/change in availability | 17 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga | Cognitive Behavioral Therapy (CBT) | Stress Education | Total
Number analyzed (Participants) | 93 | 90 | 43 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (13.3) | 35.1 (13.8) | 31.6 (13.3) | 33.1 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 62 | 29 | 158
  Male | 26 | 28 | 14 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian and Native Hawaiian or Pacific Islander | 8 | 8 | 5 | 21
  Black or African American | 3 | 5 | 3 | 11
  White | 79 | 69 | 30 | 178
  Unknown or not reported | 3 | 8 | 5 | 16
  Ethnicity: Hispanic or Latino | 11 | 6 | 1 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 93 | 90 | 43 | 226

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Treatment Response
Description: Treatment response is a dichotomous outcome coded 0=no treatment response, 1= treatment response. This treatment response coding was derived from the Clinical Global Impression-Improvement (CGI-I) measure. The CGI-I is a clinician administered instrument that assesses level of symptom change across the course of treatment. The CGI-I ranges from 1 to 7, with lower scores indicating greater improvement. Our treatment response outcome variable was coded 0 if CGI-I was 3 or more. Treatment response was coded 1 if CGI-I was rated 1 (very much improved) or 2 (much improved).
Time Frame: Biweekly from weeks 0 through 12
Measure: Number; unit: Proportion of participants
Arm/Group | Yoga | Cognitive Behavioral Therapy (CBT) | Stress Education
Number analyzed (Participants) | 93 | 90 | 43
Proportion of participants | 0.54 | 0.71 | 0.33
Statistical Analysis 1: Comparison: Yoga vs Stress Education; This comparison is from the Generalized Linear Mixed Models (GLMM) analysis using a quadratic growth curve over time. This comparison is at post-treatment. Note, although all 3 groups are included in the GLMM, this statistical test specifically compares response rates of KY vs. SE at post-treatment; Test type: Superiority; p = .03, Generalized Linear Mixed Models; Odds Ratio (OR) = 2.46, 95% CI 2-sided [1.12 to 5.42]
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy (CBT) vs Stress Education; This comparison is from the Generalized Linear Mixed Models (GLMM) analysis using a quadratic growth curve over time. This comparison is at post-treatment. Note, although all 3 groups are included in the GLMM, this statistical test specifically compares response rates of CBT vs. SE at post-treatment; Test type: Superiority; p < .001, Generalized Linear Mixed Models; Odds Ratio, log = 5, 95% CI 2-sided [2.12 to 11.82]
Statistical Analysis 3: Comparison: Yoga vs Cognitive Behavioral Therapy (CBT); This comparison is from the Generalized Linear Mixed Models (GLMM) analysis using a quadratic growth curve over time. This comparison is at post-treatment. Note, although all 3 groups are included in the GLMM, this statistical test specifically compares response rates of KY vs. CBT at post-treatment; Test type: Superiority; p = 0.07, Generalized Linear Mixed Models; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.24 to 1.03]

2. Secondary Outcome: Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A)
Time Frame: Weeks 0, 6 , 12 and 6 month follow up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 37 weeks
Description: Adverse events assessed 1x/week from baseline to 6 month follow up
Arm/Group | Yoga | Cognitive Behavioral Therapy (CBT) | Stress Education
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/90 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/93 | 1/90 | 0/43
Other Adverse Events (participants affected / at risk) | 40/93 | 34/90 | 8/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga (N=93) | Cognitive Behavioral Therapy (CBT) (N=90) | Stress Education (N=43)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga (N=93) | Cognitive Behavioral Therapy (CBT) (N=90) | Stress Education (N=43)
Amenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 16 (16) | 9 (9) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (2)
Headache (General disorders) | 1 (1) | 2 (2) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 6 (6) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Joint Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 1 (1)
Mental Distress (Psychiatric disorders) | 4 (4) | 3 (3) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nightmares (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Tingling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Vision Abnormal (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Assault (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bulimia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Faint (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flu (General disorders) | 0 (0) | 2 (2) | 0 (0)
Lymph Nodes Enlarged (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
pain (General disorders) | 0 (0) | 3 (3) | 1 (1)
Mood Change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT01912287/Prot_SAP_ICF_000.pdf